CLINICAL TRIAL: NCT01626196
Title: Multicentre, Observational, Prospective Study, Conducted on Italian Out-patients Undergoing Colonoscopy, for the Evaluation of the Main Determinants of the Patient's Acceptability of Bowel Cleansing Procedure, and of the Success of Bowel Cleansing and Caecal Intubation
Brief Title: Evaluation of the Main Determinants of Patient Acceptability of the Bowel Cleansing Procedure, and of Success of Bowel Cleansing and Caecal Intubation
Status: Completed | Type: Observational
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Other Study IDs: NIT MOV 1002
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Routine Colonoscopy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonoscopy patients: Patients undergoing with bowel cleansing procedures according to the clinics' usual routine
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This was an observational study

SUMMARY:
Several factors are important in achieving a successful colonoscopy, including patient acceptability of the bowel cleansing procedure and the overall quality of cleansing.

This observational study has been designed to explore the main determinants of acceptability of the bowel cleansing procedure to the patient in an Italian "real life" setting. In addition, the study is to examine the determinants of quality of bowel cleansing and describe aspects of the technical performance of the colonoscopy (time to reach the caecum and adenoma detection rate).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to inclusion.
* Male and female outpatients, aged ≥ 18, treated with bowel cleansing preparation the day before undergoing routine colonoscopy at selected participating centres.

Exclusion Criteria:

* Children and adolescents aged less than 18 years. Pregnant or breastfeeding women.
* Listed contra-indications to the relevant product used for the bowel cleansing procedure.
* Patients having been submitted to a previous colonoscopy over the last five years.
* Patients who have taken laxative enemas the day preceding the colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients invited for routine colonoscopy were invited to participate in hte study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Patients acceptability of the procedure | One day

SECONDARY OUTCOMES:
Time to reach the caecum | One day
Adenoma detection rate | One day

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Instituto Clinico Humanitas
Locations (1):
- IRCCS Instituto Clinico Humanitas, Milan, Rozzano, Italy